CLINICAL TRIAL: NCT03489382
Title: The BEACON Study: Protocol for Cluster RCT of a Service to Deliver Smartphone-Assisted Problem-Solving Therapy Compared to Usual Care in Men Who Present With Intentional Self-Harm to the ED in Ontario (Protocol A)
Brief Title: The BEACON Study: Smartphone-Assisted Problem-Solving Therapy in Men Presenting to the ED With Self-Harm (Protocol A)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Change in protocol design due to COVID-19 pandemic
Sponsor: University of Ottawa (Other)
Collaborators: Ottawa Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Dr. Simon Hatcher, Scientist, University of Ottawa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CTO-0790-A
Record Dates: First submitted 2018-02-27; First posted 2018-04-05 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Intentional Self-Harm; Suicide
Keywords: self-harm; problem-solving therapy; emergency department; e-therapy; suicide prevention
MeSH Terms: conditions — Self-Injurious Behavior; Suicide; Emergencies; Suicide Prevention

STUDY DESIGN:
Intervention Model Description: Multi-Centre Cluster Randomized Controlled Trial
Who Masked: Outcomes Assessor
Masking Description: All data linkage and analyses will be conducted by statisticians who are blind to the study site allocations.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): Emergency Departments providing usual care, which includes assessment in hospital followed by placement on a wait list for psychiatric services and access to regional community resources for suicide prevention.
- Smartphone Assisted PST (Experimental): Emergency Departments providing the option to refer men who self-harm to a service that will deliver smartphone-assisted problem solving therapy.
  Interventions: Other: Smartphone Assisted PST

INTERVENTIONS:
Other: Smartphone Assisted PST — Emergency Departments randomized to the study intervention will receive:
  1. Staff education incorporated into regular teaching rounds at least twice a year about the management of self-harm in the Emergency Department. This will include the dissemination of guidelines on how to ask questions about suicide, assessment of suicide risk, the creation of a management plan and how to refer patients to local mental health resources, including the study.
  2. Written materials developed by service users for men who self-harm that outline local resources, distress centre helplines, and follow-up arrangements.
  3. The option to refer men who self-harm to a service that will deliver smartphone-assisted PST specifically designed for men.
  Arms: Smartphone Assisted PST

SUMMARY:
This study evaluates the effectiveness of a smartphone-assisted problem-solving therapy (PST) service across Emergency Departments in Ontario. A total of 25 Emergency Departments have been randomized to either usual care or the smartphone-assisted PST service intervention. The main cluster randomized controlled trial will use data collected from the Institute of Clinical Evaluative Sciences (ICES) to assess the impact of this service on suicides and re-presentations to hospital for self-harm as well as other health service use one-year post study launch.

DETAILED DESCRIPTION:
Self-harm is defined as intentional self-poisoning or self-injury, whether or not there is evidence that the act was intended to result in death. In the past, the term used was 'attempted suicide.' However, peoples' motives for harming themselves are highly variable, a person may have more than one motive and motivation is hard to assess. In line with usual public policy in health and social care, the investigators use the term 'self-harm' describing a behaviour - avoiding the word 'deliberate' because many service users or consumers dislike its connotations.

In Ontario, the number of people who present to hospital emergency departments with self-harm is difficult to accurately assess, but the best estimate is about 30,000 each year. The most common form of self-harm seen in emergency departments (around 80% of episodes) is the intentional consumption of an excess of a medicinal or toxic product, whether or not there is evidence that the act was intended to result in death. Injuries, most commonly self-cutting, form 15-20% of episodes.

Two-thirds of people attending emergency departments because of self-harm are under 35 years of age. They are high users of health and social care services. Self-harm has a strong association with suicide: 7 patients per 1000 (about 1%) die by suicide in the year after attending emergency departments with a non-fatal episode (60 times the general population risk), rising to as many as 30 patients per 1000 over the next 15 years. In a recent longitudinal study conducted at the University of Toronto, "all-cause mortality following a first episode of self-poisoning was 1107 per 100,000 person-years… [with] nearly half of all deaths being suicides, accidents or undetermined intent." About a quarter of suicides are preceded by a hospital visit due to non-fatal self-harm in the previous year. It is the major identifiable risk factor for suicide. Mortality from non-suicidal causes is also high, with significantly more than the expected numbers of deaths from natural causes and from accidents. Whilst four of ten people who present with self-harm are men, they form nearly two thirds of suicides after an episode and are far more likely than women to die of premature death from other causes. The premature deaths are greatly over-represented among young people and the life years lost to the community are many.

Repetition of non-fatal self-harm stands at around 20% annually and is associated with much distress and many unresolved interpersonal problems. It is likely that any reduction in repetition of self-harm will be mirrored by a fall in subsequent suicides. The Canadian Association for Suicide Prevention blueprint for a National Suicide Prevention Strategy (CASP) has identified those who have presented to hospital with non-fatal self-harm as a high risk target group to reduce suicide.

People attending emergency departments after self-harm receive a variable standard of care in Ontario. Many are not assessed for psychological needs, and the little psychological therapy available is not usually covered by Ontario Health Insurance (OHIP). Local data from hospitals in Ottawa show that only 4 out of 10 men who present with intentional self-harm are seen by a mental health professional. Few are offered an evidence-based treatment aimed at reducing their risk of suicide or repeated self-harm. At present, assessment for self-harm in adults in Ontario is highly variable and there is no standard protocol for therapy. Assessment of suicide risk is currently a Required Operating Practice for Canadian Hospital accreditation; however, individuals identified as at-risk for suicide rarely receive recommended care.

Specialist services offer intensive and lengthy treatment for the minority of people who self-harm diagnosed with personality disorders, such as dialectical behavior therapy or mindfulness based therapy. The evidence for the effectiveness of these specialist therapies comes almost entirely from studies in women.

The investigators have received funding for a multicentre cluster randomized trial from the Ontario Strategy for Patient Oriented Research (SPOR) Support for People and Patient Oriented Research and Trials (SUPPORT) Unit funded by Canadian Institutes for Health Research (CIHR), the Ontario Ministry of Health and Long-Terms Care (MOHLTC), and the Ontario Ministry of Research, Innovation and Science (MRIS), comparing the delivery of smart phone assisted problem solving therapy with treatment as usual in men who present with self-harm. The rationale for focusing on men is that most suicides are in men and previous trials have found that providing generic treatments to everyone does not work. The intervention will build on previous work by trying to extend the range and intensity of therapy. The investigators will do this by supplementing it with a sophisticated smart phone application that has already demonstrated its effectiveness in men with substance abuse disorders. The investigators will be offering an intervention specifically designed for men who self-harm, as they are hard to engage and are more likely than women to have substance abuse problems.

Given the complexity of the proposed study, the investigators have separated the overarching research proposal into two parts, designated "Protocol A" and "Protocol B." Protocol A refers to a comprehensive secondary analysis the investigators will be carrying out using data from the Institute for Clinical Evaluative Sciences (ICES), and Protocol B refers to the active components of the intervention, those carried out with human subjects receiving six sessions of blended, problem solving therapy as opposed to routine care. The following description outlines the research protocol developed under the heading "Protocol A."

Data collected from the ICES will be used to assess the impact of our intervention on suicides and re-presentations to hospital for self-harm, as well as providing an estimation of the intervention's economic impact on the Ontario healthcare system. This data is routinely collected and housed by ICES, and access to all outcome data has been agreed upon in advance of the study launch. Given that this component of the study focuses on the evaluation of the intervention based on routinely collected population-level data, there will be no individual participant recruitment; instead, the unit of analysis will be the individual patient, with eligibility determined by the patient's presentation at either an intervention or control site's Emergency Department for self-harm. To minimize the risk of imbalances between the study arms, allocation of a site to an intervention or control arm was completed using covariate constrained allocation, based on geographic and catchment area, the availability of onsite psychiatric services assessing Emergency Department visitors, rates of representation for self-harm, and facility size, defined by the average number of presentations for self-harm over a three year period. Dichotomous primary and secondary outcome measures will be compared according to study arm, using frequencies and percentages.

The main study outcome measure for Protocol A consists of a composite measure, combining the incidence of suicide and/or representations to any Emergency Department in Ontario for self-harm in the year following the index episode of self-harm. Secondary objectives include: representation to any Emergency Department in Ontario for any reason, admission to any hospital in Ontario for any reason, hospital appointments in Ontario for any reason, primary care appointments in Ontario for any reason, mortality for reasons other than suicide, total healthcare costs, physician healthcare costs, Emergency Department health care costs, hospitalization healthcare costs, and other healthcare costs. All economic analyses will be similarly carried out with the province of Ontario considered as the population of interest. The primary composite outcome measure will be compared between the intervention and control sites using generalized linear mixed effect regression, accounting for the pre-and post-intervention measures using repeated cross-sectional analysis. Differences between the arms will be expressed as absolute and relative differences in proportions together with 95% confidence intervals. Models will account for clustering at the level of the Emergency Department and over time using random effects. Additional analyses will adjust for individual prognostic variable including age, ethnicity, pre-specified comorbidities, and repeat as compared to first-time presentations for self-harm.

The investigators will conduct a cost-utility analysis from a health system's perspective using a decision analytic model. Costs associated with the intervention will be summarized over a one-year period using a micro-costing technique. This will involve identifying, costing and valuing all resources used. An incremental cost per one additional quality-adjusted life year (QALY) gained will be estimated using one-way and probabilistic sensitivity analyses. This cost-utility analysis will adhere to the best practices for conducting and reporting of health economic evaluations.

ELIGIBILITY:
Inclusion Criteria:

* Patient has presented with an index episode of intentional self-harm at an eligible Emergency Department in Ontario, Canada.
* Patient is biologically male.
* Patient is 18 years of age or older.
* Patient has a valid OHIP number.

Exclusion Criteria:

* Patient has presented to the Emergency Department for a reason other than intentional self-harm at an eligible Emergency Department in Ontario, Canada.
* Patient is biologically female.
* Patient is under 18 years of age.
* Patient does not have a valid OHIP number.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-03 (Estimated); Primary Completion 2020-10-31 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
Change in Number of Deaths by Suicide and/or Re-Presentations to Any Emergency Department (ED) in Ontario for Self-Harm - Data from the Institute for Clinical Evaluative Sciences (ICES) | Baseline; 12 Months.
  The total number of documented suicides and/or re-presentations to any Ontario ED for self-harm will be captured by means of routinely collected administrative health data. For total number of suicides the Vital Statistics - Death database will be used. The incidence of suicide will be measured using codes drawn from the International Classification of Disease - Clinical Modification (10th edition). For the total number of re-presentations to any ED in Ontario the National Ambulatory Care Reporting System (NACRS) database will be used. Re-presentations to any ED for self-harm will also be measured using the same coding system. These numbers will be combined into a single measure, providing us with the proportion of ED visits resulting in a death by suicide or representation to an ED for self-harm, as compared to the total number of ED visits occurring at an intervention or control site. Proportions for each site will be compared to a measure taken 12 months after baseline.

SECONDARY OUTCOMES:
Change in the Number of Deaths by Suicide at a Study Site | Baseline; 12 Months.
  The total number of documented suicides will be captured for each study site by means of routinely collected administrative health data obtained from the Institute for Clinical Evaluative Sciences (ICES) using the Vital Statistics - Death database. The incidence of suicide will be measured using codes drawn from the International Classification of Disease - Clinical Modification (10th edition), and then compared against the total number of documented suicides for each study site 12 months later.
Change in Number of Re-Presentations to Any Emergency Department for Self-Harm | Baseline; 12 Months.
  The total number of documented re-presentations to any Emergency Department in Ontario for self-harm will be captured by means of routinely collected administrative health data obtained from the Institute for Clinical Evaluative Sciences (ICES) using the National Ambulatory Care Reporting System (NACRS) database. The incidence of re-presentations to any Emergency Department in Ontario for self-harm will be measured using codes drawn from the International Classification of Disease - Clinical Modification (10th edition). This measure will be compared against the total number of re-presentations to any Emergency Department in Ontario for self-harm, as measured 12 months after baseline.
Change in Number of Re-Presentations to Any Emergency Department for Any Reason | Baseline; 12 Months.
  The total number of documented re-presentations to any Emergency Department in Ontario for any reason will be captured by means of routinely collected administrative health data obtained from the Institute for Clinical Evaluative Sciences (ICES) using the National Ambulatory Care Reporting System (NACRS) database. The incidence of re-presentations to any Emergency Department in Ontario for any reason will be measured using codes drawn from the International Classification of Disease - Clinical Modification (10th edition). This measure will be compared against the total number of re-presentations to any Emergency Department in Ontario for self-harm, as measured 12 months after baseline.
Change in Number of Admissions to Any Hospital in Ontario for Any Reason | Baseline; 12 Months.
  The total number of documented presentations to any hospital in Ontario for any reason will be captured by means of routinely collected administrative health data obtained from the Institute for Clinical Evaluative Sciences (ICES) using the National Ambulatory Care Reporting System (NACRS) database. This number will be compared against the total number of admissions to any hospital in Ontario for any reason, as measured 12 months after baseline.
Change in Number of Hospital Outpatient Appointments in Ontario for Any Reason | Baseline; 12 Months.
  The total number of documented presentations hospital outpatient appointments in Ontario for any reason will be captured by means of routinely collected administrative health data obtained from the Institute for Clinical Evaluative Sciences (ICES) using the Ontario Health Insurance Plan (OHIP) database. This number will be compared against the total number of admissions to any hospital in Ontario for any reason, as measured 12 months after baseline.
Change in Number of Primary Care Appointments | Baseline; 12 Months.
  The total number of documented primary care appointments in Ontario will be captured by means of routinely collected administrative health data obtained from the Institute for Clinical Evaluative Sciences (ICES) using the Ontario Health Insurance Plan (OHIP) database. This number will be compared against the total number of primary care appointments in Ontario, as measured 12 months after baseline.
Change in Total Number of Deaths for Reasons Other Than Suicide | Baseline; 12 Months.
  The total number of documented deaths for reasons other than suicide in Ontario will be captured by means of routinely collected administrative health data obtained from the Institute for Clinical Evaluative Sciences (ICES) using the Office of the Registrar General - Deaths (ORGD) database. This number will be compared against the total number of deaths for reasons other than suicide in Ontario, as measured 12 months after baseline.
Change in Total Ontario Health Care Costs - Micro-Costing Analysis of Health-Care Resources Used in Treating Self-Harm and Suicide | Baseline; 12 Months.
  Changes in total health care costs used to treat self-harm and suicide in Ontario will be captured by means of data obtained from ICES databases. Databases: Ontario Health Insurance Plan; Discharge Abstract Database; National Ambulatory Care Reporting System; National Rehabilitation Reporting System; Continuing Care Reporting System; Ontario Mental Health Reporting System; Ontario Drug Benefit Claims; and the Assistive Devices Program. Resource costs assessed will include: physician visits, inpatient hospital admissions, home care and rehabilitation claims, use of laboratory services, and prescription drug claims for those with high drug costs as compared to income. Total costs for the intervention will also be assessed. This will include costs for training, data plans, materials, and costs associated with health care use over the one-year period. A one-year time horizon will be adopted in a base case analysis, and a lifetime horizon will be used in a scenario analysis.
Change in Ontario Physician Health Care Costs - Micro-Costing Analysis of Physician Health-Care Costs in Treating Self-Harm and Suicide | Baseline; 12 Months.
  Changes in physician health care costs in Ontario for treating self-harm and suicide in Ontario will be captured by means of routinely collected administrative health data obtained from the Institute for Clinical Evaluative Sciences (ICES) using the Ontario Health Insurance Plan (OHIP) Claims Database. This analysis will examine the cost of primary care and specialist consultations for treating self-harm and suicide in Ontario. Cost comparisons will adopt a one-year time horizon for a base case analysis, and a lifetime horizon for a scenario analysis.
Change in Ontario Emergency Department Health Care Costs | Baseline; 12 Months.
  Changes in Emergency Department health care costs in Ontario for treating self-harm and suicide will be captured by means of routinely collected administrative health data obtained from the Institute for Clinical Evaluative Sciences (ICES) using the National Ambulatory Care Reporting System (NACRS) database. This analysis will examine the cost of Ontario Emergency Department health care costs for treating self-harm and suicide. Cost comparisons will adopt a one-year time horizon for a base case analysis, and a lifetime horizon for a scenario analysis.
Change in Ontario Hospitalization Health Care Costs | Baseline; 12 Months.
  Changes in hospitalization health care costs in Ontario for treating self-harm and suicide will be captured by means of routinely collected administrative health data obtained from the Institute for Clinical Evaluative Sciences (ICES) using the Discharge Abstract Database (DAD). This analysis will examine the cost of hospitalizations for treating self-harm and suicide in Ontario, including services provided by mental health institutions, and those provided during emergency and ambulatory care visits. Cost comparisons will adopt a one-year time horizon for a base case analysis, and a lifetime horizon for a scenario analysis.
Change in Other Ontario Health Care Costs | Baseline; 12 Months.
  Other Ontario health care costs will be captured by means of routinely collected administrative health data obtained from the Institute for Clinical Evaluative Sciences (ICES) using the following databases: National Rehabilitation Reporting System (NRS); Continuing Care Reporting System (CCRS); Ontario Mental Health Reporting System (OMHRS); Ontario Drug Benefit Claims (ODB); and the Assistive Devices Program (ADP). This analysis will examine the other Ontario health care costs accrued in the treatment of self-harm and suicide, specifically the cost of home care and rehabilitation claims, cost of laboratory services, and prescription drug claims for those with high drug costs compared to income. Cost comparisons will adopt a one-year time horizon for a base case analysis, and a lifetime horizon for a scenario analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Simon Hatcher, MD, Principal Investigator — University of Ottawa; Marnin Heisel, PhD, Principal Investigator — University of Western Ontario, Canada
Locations (1):
- The Ottawa Hospital - General Campus, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Klonsky ED. Non-suicidal self-injury in United States adults: prevalence, sociodemographics, topography and functions. Psychol Med. 2011 Sep;41(9):1981-6. doi: 10.1017/S0033291710002497. Epub 2011 Jan 5. PMID 21208494
- [Background] Self-Injury Hospitalizations Details for Ontario [Internet]. Ottawa (ON): The Canadian Institute for Health Information. c2018 - [cited 2017 Feb 20] Available from: https://yourhealthsystem.cihi.ca/hsp/indepth?lang=en#/indicator/042/2/C5001/
- [Background] Bethell J, Rhodes AE. Identifying deliberate self-harm in emergency department data. Health Rep. 2009 Jun;20(2):35-42. PMID 19728584
- [Background] Gunnell D, Bennewith O, Peters TJ, House A, Hawton K. The epidemiology and management of self-harm amongst adults in England. J Public Health (Oxf). 2005 Mar;27(1):67-73. doi: 10.1093/pubmed/fdh192. Epub 2004 Nov 25. PMID 15564277
- [Background] Hawton K, Bergen H, Casey D, Simkin S, Palmer B, Cooper J, Kapur N, Horrocks J, House A, Lilley R, Noble R, Owens D. Self-harm in England: a tale of three cities. Multicentre study of self-harm. Soc Psychiatry Psychiatr Epidemiol. 2007 Jul;42(7):513-21. doi: 10.1007/s00127-007-0199-7. Epub 2007 May 21. PMID 17516016
- [Background] Health Indicators 2013 [Internet]. Ottawa (ON): The Canadian Institute for Health Information. c2013 - [cited 2017 Feb 20] Available from: https://secure.cihi.ca/free_products/HI2013_EN.pdf
- [Background] Heisel MJ, Duberstein PR. Working sensitively and effectively to reduce suicide risk among older adults. In: Kleespies PM, editor. The Oxford handbook of behavioural emergencies and crises. Oxford: Oxford University Press; 2016. P. 335-359.
- [Background] Carroll R, Metcalfe C, Gunnell D. Hospital presenting self-harm and risk of fatal and non-fatal repetition: systematic review and meta-analysis. PLoS One. 2014 Feb 28;9(2):e89944. doi: 10.1371/journal.pone.0089944. eCollection 2014. PMID 24587141
- [Background] Finkelstein Y, Macdonald EM, Hollands S, Sivilotti ML, Hutson JR, Mamdani MM, Koren G, Juurlink DN; Canadian Drug Safety and Effectiveness Research Network (CDSERN). Risk of Suicide Following Deliberate Self-poisoning. JAMA Psychiatry. 2015 Jun;72(6):570-5. doi: 10.1001/jamapsychiatry.2014.3188. PMID 25830811
- [Background] Owens D, House A. General hospital services for deliberate self-harm. Haphazard clinical provision, little research, no central strategy. J R Coll Physicians Lond. 1994 Jul-Aug;28(4):370-1. No abstract available. PMID 7965981
- [Background] Da Cruz D, Pearson A, Saini P, Miles C, While D, Swinson N, Williams A, Shaw J, Appleby L, Kapur N. Emergency department contact prior to suicide in mental health patients. Emerg Med J. 2011 Jun;28(6):467-71. doi: 10.1136/emj.2009.081869. Epub 2010 Jul 26. PMID 20660941
- [Background] Bergmans Y, Bolton MJ, Hill A, editors. The CASP blueprint for a Canadian national suicide prevention strategy [Internet]. Winnipeg, MB: Canadian Association for Suicide Prevention; 2009 [cited 2017 Feb 20]. Available: https://suicideprevention.ca/wp-content/uploads/2016/09/SuicidePreventionBlueprint0909.pdf
- [Background] Hawton K, Harriss L, Zahl D. Deaths from all causes in a long-term follow-up study of 11,583 deliberate self-harm patients. Psychol Med. 2006 Mar;36(3):397-405. doi: 10.1017/S0033291705006914. Epub 2006 Jan 10. PMID 16403244
- [Background] Comtois KA, Russo J, Snowden M, Srebnik D, Ries R, Roy-Byrne P. Factors associated with high use of public mental health services by persons with borderline personality disorder. Psychiatr Serv. 2003 Aug;54(8):1149-54. doi: 10.1176/appi.ps.54.8.1149. PMID 12883144
- [Background] Owens D, Horrocks J, House A. Fatal and non-fatal repetition of self-harm. Systematic review. Br J Psychiatry. 2002 Sep;181:193-9. doi: 10.1192/bjp.181.3.193. PMID 12204922
- [Background] Milnes D, Owens D, Blenkiron P. Problems reported by self-harm patients: perception, hopelessness, and suicidal intent. J Psychosom Res. 2002 Sep;53(3):819-22. doi: 10.1016/s0022-3999(02)00327-6. PMID 12217457
- [Background] Statistics Canada. Canadian coroner and medical examiner database: Annual report (82-214-X) [Internet]. Ottawa: Public Health Agency of Canada; c2012 [cited 2017 May 12] Available from: www.statcan.gc.ca/pub/82-214-x/82-214-x2012001-eng.pdf
- [Background] Ness J, Hawton K, Bergen H, Cooper J, Steeg S, Kapur N, Clarke M, Waters K. Alcohol use and misuse, self-harm and subsequent mortality: an epidemiological and longitudinal study from the multicentre study of self-harm in England. Emerg Med J. 2015 Oct;32(10):793-9. doi: 10.1136/emermed-2013-202753. Epub 2015 Jan 6. PMID 25564479
- [Background] Public Health Agency for Northern Ireland. Northern Ireland registry of self-harm western area: Six year summary report 2007-2012 [Internet]. Belfast: Public Health Agency; c2015 [cited February 20 2017] Available from: http://www.publichealth.hscni.net/sites/default/files/Western%20Trust%206-Year%20Report_0.pdf
- [Background] Health Canada. Acting on what we know: Preventing youth suicide in First Nations. [Internet]. Ottawa: Government of Canada; c2010 [cited 2017 December 01] Available from: http://www.hc-sc.gc.ca/fniah-spnia/pubs/promotion/_suicide/prev_youth-jeunes/index-eng.php#tphp
- [Background] Hawton K, Witt KG, Taylor Salisbury TL, Arensman E, Gunnell D, Hazell P, Townsend E, van Heeringen K. Psychosocial interventions for self-harm in adults. Cochrane Database Syst Rev. 2016 May 12;2016(5):CD012189. doi: 10.1002/14651858.CD012189. PMID 27168519
- [Background] Gustafson DH, McTavish FM, Chih MY, Atwood AK, Johnson RA, Boyle MG, Levy MS, Driscoll H, Chisholm SM, Dillenburg L, Isham A, Shah D. A smartphone application to support recovery from alcoholism: a randomized clinical trial. JAMA Psychiatry. 2014 May;71(5):566-72. doi: 10.1001/jamapsychiatry.2013.4642. PMID 24671165
- [Background] Haw C, Hawton K, Casey D, Bale E, Shepherd A. Alcohol dependence, excessive drinking and deliberate self-harm: trends and patterns in Oxford, 1989-2002. Soc Psychiatry Psychiatr Epidemiol. 2005 Dec;40(12):964-71. doi: 10.1007/s00127-005-0981-3. Epub 2005 Dec 9. PMID 16341616
- [Background] O'Connor E, Gaynes B, Burda BU, Williams C, Whitlock EP. Screening for Suicide Risk in Primary Care: A Systematic Evidence Review for the U.S. Preventive Services Task Force [Internet]. Rockville (MD): Agency for Healthcare Research and Quality (US); 2013 Apr. Report No.: 13-05188-EF-1. Available from http://www.ncbi.nlm.nih.gov/books/NBK137737/ PMID 23678511
- [Background] ICD-10-CM: International classification of diseases, 10th revision, clinical modification [Internet]. Atlanta (GA): Center for Disease Control National Center for Health Statistics. C2016 - [cited 2017 May 11] Available from: https:www.cdc.gov/nchs/icd/icd10cm.htm
- [Background] Krieger T, Meyer B, Sude K, Urech A, Maercker A, Berger T. Evaluating an e-mental health program ("deprexis") as adjunctive treatment tool in psychotherapy for depression: design of a pragmatic randomized controlled trial. BMC Psychiatry. 2014 Oct 8;14:285. doi: 10.1186/s12888-014-0285-9. PMID 25298158
- [Background] Kooistra LC, Wiersma JE, Ruwaard J, van Oppen P, Smit F, Lokkerbol J, Cuijpers P, Riper H. Blended vs. face-to-face cognitive behavioural treatment for major depression in specialized mental health care: study protocol of a randomized controlled cost-effectiveness trial. BMC Psychiatry. 2014 Oct 18;14:290. doi: 10.1186/s12888-014-0290-z. PMID 25326035
- [Background] Thompson SC, Schlehofer MM. The many sides of control motivation for high, low and illusory control. Shah JY, Gardner WL, editors. Handbook of motivation science. New York: Guilford Press; 2008, pp 41-56.
- [Background] Wright JH, Wright AS, Albano AM, Basco MR, Goldsmith LJ, Raffield T, Otto MW. Computer-assisted cognitive therapy for depression: maintaining efficacy while reducing therapist time. Am J Psychiatry. 2005 Jun;162(6):1158-64. doi: 10.1176/appi.ajp.162.6.1158. PMID 15930065
- [Background] Kleiboer A, Smit J, Bosmans J, Ruwaard J, Andersson G, Topooco N, Berger T, Krieger T, Botella C, Banos R, Chevreul K, Araya R, Cerga-Pashoja A, Cieslak R, Rogala A, Vis C, Draisma S, van Schaik A, Kemmeren L, Ebert D, Berking M, Funk B, Cuijpers P, Riper H. European COMPARative Effectiveness research on blended Depression treatment versus treatment-as-usual (E-COMPARED): study protocol for a randomized controlled, non-inferiority trial in eight European countries. Trials. 2016 Aug 3;17(1):387. doi: 10.1186/s13063-016-1511-1. PMID 27488181
- [Background] Reid SC, Kauer SD, Hearps SJ, Crooke AH, Khor AS, Sanci LA, Patton GC. A mobile phone application for the assessment and management of youth mental health problems in primary care: a randomised controlled trial. BMC Fam Pract. 2011 Nov 29;12:131. doi: 10.1186/1471-2296-12-131. PMID 22123031
- [Background] Proudfoot J, Parker G, Hadzi Pavlovic D, Manicavasagar V, Adler E, Whitton A. Community attitudes to the appropriation of mobile phones for monitoring and managing depression, anxiety, and stress. J Med Internet Res. 2010 Dec 19;12(5):e64. doi: 10.2196/jmir.1475. PMID 21169174
- [Background] Cooper J, Steeg S, Bennewith O, Lowe M, Gunnell D, House A, Hawton K, Kapur N. Are hospital services for self-harm getting better? An observational study examining management, service provision and temporal trends in England. BMJ Open. 2013 Nov 19;3(11):e003444. doi: 10.1136/bmjopen-2013-003444. PMID 24253029
- [Background] Olfson M, Marcus SC, Bridge JA. Emergency treatment of deliberate self-harm. Arch Gen Psychiatry. 2012 Jan;69(1):80-8. doi: 10.1001/archgenpsychiatry.2011.108. Epub 2011 Sep 5. PMID 21893643
- [Background] Hickey L, Hawton K, Fagg J, Weitzel H. Deliberate self-harm patients who leave the accident and emergency department without a psychiatric assessment: a neglected population at risk of suicide. J Psychosom Res. 2001 Feb;50(2):87-93. doi: 10.1016/s0022-3999(00)00225-7. PMID 11274665
- [Background] Schull M, Vermeulen T, Stukel T, Fisher E. Follow-up and shared care following discharge from the Emergency Department for exacerbations of chronic disease. Can J Emerg Med. 2013; 13(Suppl 1):LOP05
- [Background] Schoen C, Osborn R, Squires D, Doty M, Rasmussen P, Pierson R, Applebaum S. A survey of primary care doctors in ten countries shows progress in use of health information technology, less in other areas. Health Aff (Millwood). 2012 Dec;31(12):2805-16. doi: 10.1377/hlthaff.2012.0884. Epub 2012 Nov 15. PMID 23154997
- [Background] Tyrer P, Thompson S, Schmidt U, Jones V, Knapp M, Davidson K, Catalan J, Airlie J, Baxter S, Byford S, Byrne G, Cameron S, Caplan R, Cooper S, Ferguson B, Freeman C, Frost S, Godley J, Greenshields J, Henderson J, Holden N, Keech P, Kim L, Logan K, Manley C, MacLeod A, Murphy R, Patience L, Ramsay L, De Munroz S, Scott J, Seivewright H, Sivakumar K, Tata P, Thornton S, Ukoumunne OC, Wessely S. Randomized controlled trial of brief cognitive behaviour therapy versus treatment as usual in recurrent deliberate self-harm: the POPMACT study. Psychol Med. 2003 Aug;33(6):969-76. doi: 10.1017/s0033291703008171. PMID 12946081
- [Background] Hatcher S, Sharon C, Parag V, Collins N. Problem-solving therapy for people who present to hospital with self-harm: Zelen randomised controlled trial. Br J Psychiatry. 2011 Oct;199(4):310-6. doi: 10.1192/bjp.bp.110.090126. Epub 2011 Aug 4. PMID 21816868
- [Background] Akbari A, Mayhew A, Al-Alawi MA, Grimshaw J, Winkens R, Glidewell E, Pritchard C, Thomas R, Fraser C. Interventions to improve outpatient referrals from primary care to secondary care. Cochrane Database Syst Rev. 2008 Oct 8;2008(4):CD005471. doi: 10.1002/14651858.CD005471.pub2. PMID 18843691
- [Background] Suicide Prevention Resource Center. Caring for adult patients with suicide risk: A consensus guide for emergency departments [Internet]. Waltham (MA): Education Development Center Inc.; 2015 [cited 2017 Feb 20]. Available from: http://www.sprc.org/sites/default/files/EDGuide_full.pdf
- [Background] Suicide Prevention Resource Center. Preventing suicide among men in the middle years: Recommendations for suicide prevention programs [Internet]. Waltham (MA): Education Development Center Inc.; 2016 [cited 2017 Feb 20]. Available from: http://www.sprc.org/sites/default/files/resource-program/SPRC_MiMYReportFinal_0.pdf
- [Background] Carroll R, Metcalfe C, Gunnell D. Hospital management of self-harm patients and risk of repetition: systematic review and meta-analysis. J Affect Disord. 2014 Oct;168:476-83. doi: 10.1016/j.jad.2014.06.027. Epub 2014 Jun 21. PMID 25128754
- [Background] Canadian Coalition for Seniors' Mental Health. National guidelines for seniors' mental health: The assessment of suicide risk and prevention of suicide. [Internet] Toronto: Canadian Coalition for Seniors' Mental Health; c2006 [cited 2017 Feb 20] Available from: https://ccsmh.ca/wp-content/uploads/2016/03/NatlGuideline_Suicide.pdf
- [Background] Andreasson K, Krogh J, Rosenbaum B, Gluud C, Jobes DA, Nordentoft M. The DiaS trial: dialectical behavior therapy versus collaborative assessment and management of suicidality on self-harm in patients with a recent suicide attempt and borderline personality disorder traits - study protocol for a randomized controlled trial. Trials. 2014 May 29;15:194. doi: 10.1186/1745-6215-15-194. PMID 24885904
- [Background] Andreasson K, Krogh J, Wenneberg C, Jessen HK, Krakauer K, Gluud C, Thomsen RR, Randers L, Nordentoft M. EFFECTIVENESS OF DIALECTICAL BEHAVIOR THERAPY VERSUS COLLABORATIVE ASSESSMENT AND MANAGEMENT OF SUICIDALITY TREATMENT FOR REDUCTION OF SELF-HARM IN ADULTS WITH BORDERLINE PERSONALITY TRAITS AND DISORDER-A RANDOMIZED OBSERVER-BLINDED CLINICAL TRIAL. Depress Anxiety. 2016 Jun;33(6):520-30. doi: 10.1002/da.22472. Epub 2016 Feb 8. PMID 26854478
- [Background] Morthorst B, Krogh J, Erlangsen A, Alberdi F, Nordentoft M. Effect of assertive outreach after suicide attempt in the AID (assertive intervention for deliberate self harm) trial: randomised controlled trial. BMJ. 2012 Aug 22;345:e4972. doi: 10.1136/bmj.e4972. PMID 22915730
- [Background] Moulton LH. Covariate-based constrained randomization of group-randomized trials. Clin Trials. 2004;1(3):297-305. doi: 10.1191/1740774504cn024oa. PMID 16279255
- [Background] Ukoumunne OC, Thompson SG. Analysis of cluster randomized trials with repeated cross-sectional binary measurements. Stat Med. 2001 Feb 15;20(3):417-33. doi: 10.1002/1097-0258(20010215)20:33.0.co;2-g. PMID 11180311
- [Background] Gold MR, Seigel JE, Russell LB, Weinstein MC, editors. Cost-effectiveness in health and medicine. New York: Oxford University Press; 1996.
- [Background] Canadian Agency for Drugs and Technologies in Health. Guidelines for the economic evaluation of health technologies. 4th Ed. [Internet]. Ottawa: Canadian Agency for Drugs and Technologies in Health; c2017 [cited 2017 May 11] Available from: https://www.cadth.ca/guidelines-economic-evaluation-health-technologies-canada-4th-edition
- [Background] Husereau D, Drummond M, Petrou S, Carswell C, Moher D, Greenberg D, Augustovski F, Briggs AH, Mauskopf J, Loder E; ISPOR Health Economic Evaluation Publication Guidelines-CHEERS Good Reporting Practices Task Force. Consolidated Health Economic Evaluation Reporting Standards (CHEERS)--explanation and elaboration: a report of the ISPOR Health Economic Evaluation Publication Guidelines Good Reporting Practices Task Force. Value Health. 2013 Mar-Apr;16(2):231-50. doi: 10.1016/j.jval.2013.02.002. PMID 23538175
- [Background] Campbell MK, Elbourne DR, Altman DG; CONSORT group. CONSORT statement: extension to cluster randomised trials. BMJ. 2004 Mar 20;328(7441):702-8. doi: 10.1136/bmj.328.7441.702. No abstract available. PMID 15031246
- [Background] Canadian Institutes of Health Research, Natural Science and Engineering Research Council of Canada, and Social Sciences and Humanities Research Council. Tri-council policy statement: Ethical conduct for research involving humans. [Internet] Ottawa: Government of Canada; c2014 [cited 2017 May 11] Available from: www.pre.ethics.gc.ca/pdf/eng/tcps2-2014/TCPS_2_FINAL_Web.pdf
- [Background] Schaffer A, Sinyor M, Kurdyak P, Vigod S, Sareen J, Reis C, Green D, Bolton J, Rhodes A, Grigoriadis S, Cairney J, Cheung A. Population-based analysis of health care contacts among suicide decedents: identifying opportunities for more targeted suicide prevention strategies. World Psychiatry. 2016 Jun;15(2):135-45. doi: 10.1002/wps.20321. PMID 27265704
- [Derived] Witt KG, Hetrick SE, Rajaram G, Hazell P, Taylor Salisbury TL, Townsend E, Hawton K. Psychosocial interventions for self-harm in adults. Cochrane Database Syst Rev. 2021 Apr 22;4(4):CD013668. doi: 10.1002/14651858.CD013668.pub2. PMID 33884617

DOCUMENTS (1):
  • Study Protocol (2017-12-01): https://cdn.clinicaltrials.gov/large-docs/82/NCT03489382/Prot_000.pdf